CLINICAL TRIAL: NCT04890626
Title: Randomized Clinical Trial to Evaluate the Efficacy of Different Treatments in Patients With COVID-19
Brief Title: Clinical Trial to Evaluate the Efficacy of Different Treatments in Patients With COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PanCOVID
Record Dates: First submitted 2021-05-17; First posted 2021-05-18 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; baricitinib; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Main randomization. Patients will be randomized to Emtricitabine / Tenofovir disoproxil fumarate or no treatment.
  Rescue randomization: patients with oxygen requirements, O2 Sat <95% at any time, and at least one of the following inflammation markers: IL-6, CRP, D-dimer, LDH or ferritin above the upper limit of the normal range. Arms:
  * dexamethasone + Baricitinib
  * dexamethasone
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Main randomization.Arm: Emtricitabine / Tenofovir disoproxil fumarate (Experimental): Emtricitabine / Tenofovir disoproxil fumarate
  Interventions: Drug: Emtricitabine/Tenofovir Disoproxil Fumarate 200 MG-245 MG Oral Tablet [TRUVADA]
- Main randomization.Arm: No treatment (No Intervention): No treatment
- Rescue randomization: Arm: Dexamethasone + Baricitinib (Other): Rescue randomization: patients with oxygen requirements, O2 Sat <95% at any time, and at least one of the following inflammation markers: IL-6, CRP, D-dimer, LDH or ferritin above the upper limit of the normal range. Arms: Dexamethasone + Baricitinib or Dexamethasone.
  Interventions: Drug: Baricitinib + dexamethasone
- Rescue randomization: Arm: Dexamethasone (Other): Rescue randomization: patients with oxygen requirements, O2 Sat <95% at any time, and at least one of the following inflammation markers: IL-6, CRP, D-dimer, LDH or ferritin above the upper limit of the normal range. Arms: Dexamethasone + Baricitinib or Dexamethasone.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Emtricitabine/Tenofovir Disoproxil Fumarate 200 MG-245 MG Oral Tablet [TRUVADA] — Main randomization
  Arms: Main randomization.Arm: Emtricitabine / Tenofovir disoproxil fumarate
Drug: Baricitinib + dexamethasone — Rescue randomization
  Arms: Rescue randomization: Arm: Dexamethasone + Baricitinib
Drug: Dexamethasone — Rescue randomization
  Arms: Rescue randomization: Arm: Dexamethasone

SUMMARY:
Currently COVID-19 is an international public health emergency. Most COVID-19 patients have mild or uncomplicated disease, but approximately 14% develop severe disease that requires hospitalization and oxygen therapy, and up to 5% of patients require admission to Intensive Care Units.

To date, the only treatments that have shown efficacy in a clinical trial are remdesivir and dexamethasone. The main objective is to provide reliable estimates on the effects of different treatment strategies on the outcome and mortality of patients with SARS-CoV-2 infection.

ELIGIBILITY:
First randomization

Inclusion criteria.

* Men and women agree to participate in the study by signing the informed consent.
* Men and women aged ≥ 60 years.
* Men and women aged ≥18 years <60 years with ≥ 2 comorbidities of the following: hypertension, obesity, diabetes, cirrhosis, chronic neurological disease, active cancer, heart failure, ischemic heart disease, COPD.
* Patient with a diagnosis of SARS-CoV-2 infection confirmed by PCR or rapid diagnostic test prior to randomization.
* Patients with symptoms and signs compatible with active infection.
* Men and women of reproductive capacity must agree to use highly effective contraceptive methods (diaphragm plus spermicide or male condom plus spermicide, oral contraceptive combined with a second method of contraceptive implant, injectable contraceptive, permanent intrauterine device, sexual abstinence or vasectomy) during your participation in the study and within 30 days of the last visit.
* In addition, women participating in the study with reproductive capacity must have a negative pregnancy test at the time of inclusion.

Exclusion criteria.

* Patients participating in any other clinical trial with drugs with potential antiviral action for SARS-CoV-2
* Concomitant treatment with drugs other than the treatments included in this study with demonstrated or potential action against SARS-CoV-2 in the 24 hours prior to the administration of the study treatment.
* Patients who are already receiving any of the study drugs.
* Patients treated with corticosteroids at immunosuppressive doses (15 mg / day in the 7 days prior to the onset of symptoms).
* Evidence of multi-organ failure.
* HIV positive, confirmed by rapid test before inclusion.
* Patients who require reservoir, mechanical ventilation or present acute respiratory distress criteria at the time of inclusion.
* ALT or AST> 5 times the upper limit of normal during screening.
* Creatinine clearance less than 60 ml / min during screening.
* Pregnancy test with positive result during screening.
* Women who are breastfeeding.
* Patients with known hypersensitivity to any of the drugs in the treatment branches of the study, their metabolites or excipients.
* Patients who receive medication incompatible with the study drugs after reviewing possible interactions.
* Patients who present any contraindication or condition that is included in the section on warnings and special precautions for the use of the technical sheets of the drugs under study (Emtricitabine / Tenofovir disoproxil, and remdesivir) or any other reason that the research team has criteria is reason. not to be included in the study.
* Subjects who are not able to understand the information sheet and are unable to sign the informed consent

Second randomization (if applicable):

Patients already included in the study and initially randomized may be re-randomized at any time if they present an O2 Sat <95% (need for oxygen therapy) and at least 1 marker of inflammation of the following: IL-6, CRP, D-Dimer , LDH, or ferritin above the upper limit of the normal range. This randomization can only be done in hospitalized patients. Patients will receive one of the following arms of treatment:

* Baricitinib and dexamethasone
* Dexamethasone

Exclusion criteria (rescue randomization):

* Non-hospitalized patient
* Being receiving cytotoxic or biological treatments (such as TNF inhibitors, anti interleukin 1, anti-interleukin 6 (tocilizumab or sarilumab), therapies against B or T cells (rituximab), interferon or Janus kinase inhibitors.
* Have ever received convalescent plasma or intravenous immunoglobulins.
* Suspicion of suffering from another serious bacterial, fungal or viral infection in addition to COVID-19 that in the opinion of the researcher could be a risk to receive the research products.
* Have received a live vaccine 4 weeks before screening
* Require mechanical ventilation or ECMO
* Patient with a history of thromboembolic disease: deep vein thrombosis and / or pulmonary embolism within 12 weeks prior to randomization or have a history of recurrent thromboembolic disease
* Neutropenia <1000 cells / μL
* Lymphopenia <200 cells / μL
* GOT or GPT> 5 times the upper limit of normal
* MDRD <30 mL / min
* History of hypersensitivity to baricitinib or its components.
* Pregnant or planning pregnancy or lactating during the study
* Are using or will be using a blood purification instrument to remove pro-inflammatory cytokines.
* A life expectancy <48 hours from screening.
* Contraindication to take the study medication or investigator criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2020-04-04 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
Mortality | at 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://pancovidtrial.net/